CLINICAL TRIAL: NCT00234897
Title: Humira Efficacy Response Optimization Study in Subjects With Active Rheumatoid Arthritis (HERO)
Brief Title: Efficacy of HUMIRA in Subjects With Active Rheumatoid Arthritis
Acronym: HERO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M04-684; HERO
Record Dates: First submitted 2005-09-13; First posted 2005-10-10 (Estimated); Last update posted 2007-08-29 (Estimated); Status verified 2007-08

CONDITIONS: Rheumatoid Arthritis
Keywords: adalimumab; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: adalimumab

SUMMARY:
The purpose of the study is to assess the efficacy of adalimumab in subjects with rheumatoid arthritis focusing on subject-reported outcomes and early response to treatment

ELIGIBILITY:
Inclusion Criteria:

* Subject was age 18 or older and in good health (Investigator discretion) with a recent stable medical history.
* Subject, based on assessment of investigator, meets the definition of active RA

Exclusion Criteria:

* Subject considered by the investigator, for any reason, to be an unsuitable candidate for the study
* Female subject who is pregnant or breast-feeding or considering becoming pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1938 (Actual)
Dates: Start 2004-08

PRIMARY OUTCOMES:
Patient reported outcomes, clinical response indicators.

SECONDARY OUTCOMES:
Subject reported assessments of disease activity, physician reported assessments of disease activity, safety parameters, clinical response indicators.

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Paperiello, Study Director — Abbott
Locations (1):
- Global Medical Information - Abbott, North Chicago, Illinois, United States